CLINICAL TRIAL: NCT07068750
Title: Evaluation of Implant Site Preparation With Three Different Drilling Systems in Posterior Maxilla (Randomized Controlled Clinical Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ALZAHRANI,MOHAMMED AHMED Y (Other)
Responsible Party: Sponsor-Investigator, ALZAHRANI,MOHAMMED AHMED Y, B.D.S (2017) Faculty of Dentistry, Mansoura University, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A01011023OM
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Evaluation of Implant Site Preparation With Three Different Drilling Systems in Posterior Maxilla

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I: 10 patients received dental implants using single drilling system in posterior maxilla (Active Comparator)
  Interventions: Procedure: patients received dental implants using single drilling system in posterior maxilla
- Group II: 10 patients received dental implants using Densah burs in posterior maxilla (Active Comparator)
  Interventions: Procedure: patients received dental implants using Densah burs in posterior maxilla
- Group III: 10 patients received dental implants using conventional drills in posterior maxilla (Active Comparator)
  Interventions: Procedure: patients received dental implants using conventional drills in posterior maxilla

INTERVENTIONS:
Procedure: patients received dental implants using single drilling system in posterior maxilla — All patients will be operated under local anaesthesia Articaine hydrochloride 4% with Epinephrine (1:100,000). Crestal incision will performed and full thickness mucoperiosteal flap will be reflected to access the site. The implant will be prepared using the new specially designed drill. These drills are available with four drilling lengths (7, 9, 11, 13 mm) characterized by different color codes, and three different diameters (4, 4.5, 5 mm). They allow a single drilling procedure before implant placement in bone with all types. Drilling speed of 1500 RPM and profuse normal saline irrigation will be used throughout the drilling procedure. Tapered implants will be inserted in all patients with insertion torque 30-50Ncm. Suturing of the flap with interrupted sutures, using 5/0 polypropylene suturing material (According to the protocol provided by the manufacturer).
  Arms: Group I: 10 patients received dental implants using single drilling system in posterior maxilla
Procedure: patients received dental implants using Densah burs in posterior maxilla — All patients will be operated under local anaesthesia Articaine hydrochloride 4% with Epinephrine (1:100,000). Crestal incision will be performed and full thickness mucoperiosteal flap will be reflected to access the site. Implant sites will be prepared using osseodensification burs (Densah, Versah) at 1200 rpm in the following sequence: (I) pilot (clockwise); (II) WT1828 (counterclockwise), and (III) WT2838 (counterclockwise). These burs have a cutting chisel edge, a tapered shank and non- cutting edges with four or more lands with a negative rake angle. Suturing of the flap with interrupted sutures, using 5/0 polypropylene suturing material (According to the protocol provided by the manufacturer).
  Arms: Group II: 10 patients received dental implants using Densah burs in posterior maxilla
Procedure: patients received dental implants using conventional drills in posterior maxilla — All patients will be operated under local anaesthesia Articaine hydrochloride 4% with Epinephrine (1:100,000). Crestal incision will be performed and full thickness mucoperiosteal flap will be reflected to access the site. Implant sites will be prepared using conventional surgical drills at 1200 rpm. Suturing of the flap with interrupted sutures, using 5/0 polypropylene suturing material (According to the protocol provided by the manufacturer).
  Arms: Group III: 10 patients received dental implants using conventional drills in posterior maxilla

SUMMARY:
The rationale for conducting this study is to compare between three implant drilling systems (conventional sequential system, single drilling system and osseodensification surgical drills) for implant site preparation in the posterior maxillay region through measuring implant stability and bone density around dental implants. Therefore, the primary objective of this study is to evaluate the primary and secondary implant stability performed by the three types through measuring implant stability quotient (ISQ), whereas the secondary objective is to assess marginal bone loss, the operation time for the osteotomy preparation, and finally bone density through measuring grey values on CBCT around implants for all drilling methods at different evaluation intervals of the study.

DETAILED DESCRIPTION:
Primary stability is a critical factor that determines the long-term success of dental implants. It is responsible for preventing the micro- motion of the implant in the bone site, promoting natural healing and effective bone formation until adequate biological stability has been established. Primary stability of dental implants is highly dependent on implant design, surgical technique and the bone density and quality. Conventional implant shaping drills are widely used because they are easy to handle, time-efficient, and not expensive. Nevertheless, the heat that they generate might cause tissue damage, necrosis to the surrounding structures, difficulty in providing a proper three-dimensional positioning and the risk of invading and injuring important anatomical structures such as the inferior alveolar nerve and the Schneiderian membrane. Hence, several studies introduce different techniques and methods to resolve these problems. Recently, new hollow drill in a single drilling system was developed. It was hypothesized that hollow drill design with single drilling system results in decreasing the time for surgery (faster implant placement) and minimum bone removal for implant site preparation. Moreover, it was found that it reduces bone trauma, micro-fractures and allow fasters healing time. Moreover, the hollow design of the single drilling system allows harvesting of the bone core, that bone which result during the osteotomy site preparation can be used in bone grafting as autogenous bone grafting material. Osseodensification (OD) is also a new method of biomechanical bone preparation performed for dental implant placement. The procedure is characterized by low plastic deformation of bone that is created by rolling and sliding contact using a densifying bur that is fluted such that it densifies the bone with minimal heat elevation. OD, a bone nonextraction technique, was developed by Huwais 2013 and done using specially designed burs (Densah™ burs) that help densify bone as they prepare an osteotomy these burs provide advantages of both osteotomes combining the speed along with improved tactile control of the drills during osteotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient between 20-50 years old.
2. remaining bone height of more than 8 mm, remaining bone width of 6 mm
3. Adequate keratinized soft tissue.
4. Favorable pattern of occlusion.
5. Good oral hygiene.
6. Patient ability to comply with the required recall visits

Exclusion Criteria:

1. Insufficient bone width (less than 6 mm) mesiodistal or buccolingually.
2. Patients having any uncontrolled systemic disease which could affect bone healing.
3. Patients treated with radiotherapy to the head and neck area within the past 12 months.
4. Heavy Smokers (more than 20 cigarette per day) according to WHO.
5. Inability or unwillingness to return for follow-up visits.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
primary and secondary implant stability | the primary stability will be taken immediately after implant placement. while secondary implant stability will be taken after 6-months
  the primary objective of this study is to evaluate the primary and secondary implant stability performed by the three types through measuring implant stability quotient (ISQ)

SECONDARY OUTCOMES:
assessment of marginal bone loss | marginal bone loss will be measured after 6 months from implant placement
  The secondary objective is to assess marginal bone loss measured on CBCT around implants for all drilling methods at different evaluation intervals of the study.
operation time | operation time will be measured immediately during implant placement in minutes.
  The secondary objective is to assess the operation time for the osteotomy preparation in each study group.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided